CLINICAL TRIAL: NCT03493087
Title: Underlying Causes of Low Vitamin K Status in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-17036789
Record Dates: First submitted 2018-02-09; First posted 2018-04-10 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Dialysis, Vitamin-K, Malnutrition
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition | interventions — Vitamin K

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menakinon-7 (Active Comparator): Menakinon-7 360 µg tablet by mouth, every day for 6 weeks
  Interventions: Dietary Supplement: Menakinon 7
- Diet with vitamin K (Active Comparator): Diet rich in vitamin K for 6 weeks
  Interventions: Dietary Supplement: Diet rich in vitamin K

INTERVENTIONS:
Dietary Supplement: Menakinon 7 — Menakinon 7 - One tablet a day against vitamin K deficiency
  Arms: Menakinon-7
Dietary Supplement: Diet rich in vitamin K — Diet with large content of vegetables and dairy products
  Arms: Diet with vitamin K

SUMMARY:
Studies have shown that patients with chronic kidney disease in hemodialysis have a low vitamin K status which is believed to be related to an increased risk of atherosclerosis and increased bleeding tendency. The underlying causes of low vitamin K status in hemodialysis patients is unknown. Thus, the aim of this study is to investigate why hemodialysis patients have a low vitamin K status and how to improve it.

This study is composed of five trials. Four of them are based on possible hypotheses to the low vitamin K status. The hypotheses are:

1. The daily intake of vitamin K is insufficient.
2. Vitamin K is removed from the blood during dialysis.
3. Absorption in the intestines is impaired.
4. The analysis method (dephosphorylated-uncarboxylated MGP) is influenced by the patients' protein intake.

The purpose of the fifth trial is to investigate solutions to improve the vitamin K status of hemodialysis. One is to improve vitamin K status through diet with an increased focus on foods with high concentrations of vitamin K while considering phosphate, potassium and fluid restrictions. The second is to increase vitamin K status through a daily supplement of 360µg Menakinon-7.

DETAILED DESCRIPTION:
Studies have reported a low vitamin K status in chronic kidney disease patients in hemodialysis linked to an increased risk of atherosclerosis and increased bleeding tendency. The overall aim of this study is to investigate the underlying causes of the reported low vitamin K status and to improve the patients' vitamin K status through diet and supplement. The study is divided in 5 sub-trials listed below. Sub-trial 1-4 focuses on determining the underlying course of low vitamin K status while sub-trial 5 deals with possible solutions to the reported low vitamin K status.

The analysis method used to determine vitamin K status is dephosphorylated-uncarboxylated Matrix-Gla-Protein (dp-ucMGP). Dp-ucMGP is the inactive form of the protein MGP whose activation is vitamin K dependent. The dp-ucMGP analysis method is not a direct measure of vitamin K status. However, an increased concentration of dp-ucMGP is a manifestation of a low vitamin K status and vice versa.

Sub-trial 1: Intake of vitamin K Aim: To assess the patients' intake of vitamin K. Hypothesis: The daily intake of vitamin K is insufficient. Method: Patients are asked to fill out a food frequency questionnaire (FFQ). The FFQ is based on their intake of different foods rich in vitamin K during the last month. To compare the results from the FFQ with their actual vitamin K status a blood sample is collected and analyzed to determine dp-ucMGP. Participants: 30.

Sub-trial 2: The influence of dialysis Aim: To examine whether vitamin K status is compromised during dialysis. Hypothesis: Vitamin K is removed from the blood during dialysis. Method: A blood test is collected before and after dialysis and analyzed to determine dp-ucMGP. At the end of the dialysis a sample of the remaining dialysis-water is collected and analyzed to determine dp-ucMGP. Furthermore, the patients will be weighed before and after dialysis with the purpose of calculating concentrations. Participants: 16 (the analysis of the dialysis water is done for five patients at first, if the results are useful the analysis is done for every participant).

Sub-trial 3: Absorption Aim: To investigate whether a decreased absorption can be the cause of the low vitamin K status. Hypothesis: Absorption in the intestines is impaired. Method: A D-xylose test is performed. The participants are given a dose of 15g D-xylose dissolved in water and after one hour a sample of blood is collected to determine D-xylose in serum. Prior to this trial the patients need to be fasting.The patients are asked to fill out a FFQ concerning their intake of fat during the last month. Participants: 16

Sub-trial 4: Concentrations of dp-ucMGP is influenced by a low protein intake. Aim: To determine if a low protein intake influence the dp-ucMGP analysis method. Hypothesis: The analysis method (dephosphorylated-uncarboxylated MGP) is influenced by the patients' protein intake. Method: Patients are given a daily protein supplement for 14 days. Before and after the intervention a blood test is collected and the concentration of dp-ucMGP is determined and compared. Moreover, the patients are asked to fill out a FFQ concerning their intake of protein during the last month. Participants: 16

Sub-trial 5: Intervention with vitamin K Aim: To investigate whether a diet or supplement with tablets is best for improve vitamin K status. Hypothesis: If the intake of vitamin K is insufficient the diet rich in vitamin K should be sufficient. However, if absorption is compromised or vitamin K is influenced by dialysis a larger dose of vitamin K might be necessary. Method: This trial lasts for 15 weeks divided in two periods of six weeks and a three week wash out period in-between. One period focuses on a diet rich in vitamin K while dealing with the possible restrictions on phosphate, potassium and fluid for hemodialysis patients. The intervention in the other period consists of a supplement of 360μg Menakinon-7/day. Blood samples are collected at the beginning, middle and end of both periods. These blood samples are analyzed to determine dp-uc-MGP during the intervention period. Moreover, coagulations factor 2, 7, 10, vitamin A and D status and calcification propency score analysis will be done as well if the funds allow it. Patients are asked to fill out a questionnaire concerning physical and mental wellbeing and the presence of bruising at the beginning and end of both periods to determine whether vitamin K has an effect. Participants: 24

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Hemodialysis (> 3 months) at Herlev Hospital, Nephrological department
* Understands and are able to read danish
* Able to collaborate on diet etc.

Exclusion Criteria:

* Warfarin treatment
* Pregnant or breastfeeding
* Prior intake of vitamin K supplements
* Short bowl disease, pancreatitis or other malabsorption diseases/syndromes
* Dementia
* Diabetes Mellitus (only an exclusion criterion in sub-trial 3: Absorption of vitamin K)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Δ-dp-uc-MGP (Sub-trial 5) | 15 weeks
  Comparison of concentration of dp-ucMGP in blood samples through out the intervention

SECONDARY OUTCOMES:
dp-ucMGP status (Sub-trial 1) | 1 day
  Concentration of dp-ucMGP in a blood sample collected before dialysis
Vitamin K intake (Sub-trial 1) | 1 month
  Intake of vitamin K is estimated from FFQ results
dp-ucMGP concentration in dialysis water (Sub-trial 2) | 1 day
  A sample of dialysis water is tested for dp-ucMGP
Δ-concentration of dp-ucMGP (Sub-trial 2) | 1 day
  Concentration of dp-ucMGP in a blood sample collected before dialysis is compared with the concentration in a blood sample collected after dialysis
Δ-weight (Sub-trial 2) | 1 day
  The patient's weight before and after dialysis is compared
Concentration of D-xylose (Sub-trial 3) | 1 day
  Concentration of D-xylose in the blood an hour after intake of 15g of D-xylose
Fat in the diet (Sub-trial 3) | 1 day
  The amount of fat in the diet is assessed from FFQ results
Δ-dp-uc-MGP (Sub-trial 4) | 14 day
  intervention with protein is compared with the concentration in a blood sample collected after the intervention
Protein in the diet (Sub-trial 4) | 14 days
  The amount of protein in the diet is assessed from FFQ results
Calcification (Sub-trial 5) | 15 weeks
  Blood samples are analyzed via calcification propensity score, T50
Quality of life (Sub-trial 5) | 15 weeks
  The results from mental and physical well being questionnaires are compared Based on SF-36 Danish version. Eight questions with scales ranges from 1-5 with 5 being the worse outcome. The questions are looked at individually and together.
The patient's perception of the presence of bruises (Sub-trial 5) | 15 weeks
  The patient assess the changes in bruising in a questionnaire.
Δ-factor 2, 7,10 concentration (Sub-trial 5) | 15 weeks
  Comparison of concentration of factor 2,7,10 in blood samples before and after both interventions

OTHER OUTCOMES:
Phosphate (Sub-trial 5) | 15 weeks
  Changes in p-phosphate through out the intervention period
Potassium (Sub-trial 5) | 15 weeks
  Changes in p-potassium through out the intervention period
Vitamin A (Sub-trial 5) | 15 weeks
  Changes in p-vitamin A through out the supplement period
Vitamin D (Sub-trial 5) | 15 weeks
  Changes in p-vitamin D through out the supplement period

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, Study Director — University of Copenhagen
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No